CLINICAL TRIAL: NCT06199414
Title: Vascular Closure With Novel External Compression Device After Atrial Fibrillation Ablation: The LockeT Study
Brief Title: Vascular Closure With Novel External Compression Device: The LockeT Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRRF_LockeT Retrospect_0020
Record Dates: First submitted 2023-12-29; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation; Hemostasis
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects with Figure-of-eight (F-8) suture: This is the group of subjects for whom Figure-of-eight (F-8) suture is used for their venous closure.
  Interventions: Device: Venous Closure
- Subjects with LockeT Device: This is the group of subjects for whom LockeT device is used for their venous closure.
  Interventions: Device: Venous Closure

INTERVENTIONS:
Device: Venous Closure — Vascular closure to achieve vascular hemostasis following femoral access with large bore sheaths in catheter ablation procedures

SUMMARY:
Single center, retrospective review study comparing Figure of Eight suture to LockeT, enrolling approximately 70 patients.

DETAILED DESCRIPTION:
The volume of catheter ablation procedures for the treatment of atrial fibrillation and other arrhythmias are on the rise in the United States and worldwide. Despite refinement in ablation tools and techniques which has led to a significant decline in complication rates, achieving vascular hemostasis following femoral access with large bore sheaths remains a challenge. Manual compression (MC) the current standard of care, requires bedrest, often up to 8 hours. This prolonged bedrest is associated with longer length of stay and at times complications from indwelling catheters.

Other methods of vascular closure include figure-of-eight (F-8) a, subcutaneous suture or Z-stitch or fellow's stitch has been evaluated as a means to achieve homeostasis following major cardiovascular procedures. One pooled meta-analysis of six studies including 982 patients demonstrated that F-8 is safe and effective means of achieving hemostasis. In comparison to MC time to hemostasis was significantly lower and overall access site complications like hematoma, bleeding was also noted to be lower in F-8 group.

In recent years, invasive, vascular closure devices have become popular. However, results continue to suggest that the risk versus benefit has not been definitively demonstrated. LockeT is a new suture retention device designed to closely mimic manual compression without the need for a healthcare professional to stand bedside.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet the following criteria to be included in this study.

* Subjects must be at least 18 years of age.
* Subjects underwent Atrial Fibrillation radiofrequency ablation procedure.
* Subjects must have undergone F-8 or LockeT for venous closure.

Exclusion Criteria:

If a subject meet any of the following criteria will be excluded from study participation.

* Subjects under the age of 18.
* Subject's electrophysiology procedure is not planned to access the left atrium or ventricle.
* Subjects in which F-8 or a LockeT was not used.
* If the EP physician detected a formed hematoma prior to venous closure, that patient will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include who underwent AF ablation and required F-8 or LockeT post procedure.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of LockeT device - Time to no oozing/hemostasis | 1 week
  To assess the effectiveness of using LockeT to retain sutures and pressure to gain hemostasis after venous procedures.
  Time to no oozing/hemostasis (mins/hours)
Effectiveness of LockeT device - Time to Ambulate | 1 week
  To assess the effectiveness of using LockeT to retain sutures and pressure to gain hemostasis after venous procedures.
  Time to no oozing/hemostasis (mins/hours)

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (2):
- United States (2):
  - Kansas City Heart Rhythm Institute - Roe Clinic, Overland Park, Kansas
  - Overland Park Regional Medical Center, Overland Park, Kansas

REFERENCES:
- [Background] Natale A, Mohanty S, Liu PY, Mittal S, Al-Ahmad A, De Lurgio DB, Horton R, Spear W, Bailey S, Bunch J, Musat D, O'Neill P, Compton S, Turakhia MP; AMBULATE Trial Investigators. Venous Vascular Closure System Versus Manual Compression Following Multiple Access Electrophysiology Procedures: The AMBULATE Trial. JACC Clin Electrophysiol. 2020 Jan;6(1):111-124. doi: 10.1016/j.jacep.2019.08.013. Epub 2019 Oct 30. PMID 31971899
- [Background] Mujer MT, Al-Abcha A, Flores J, Saleh Y, Robinson P. A comparison of figure-of-8-suture versus manual compression for venous access closure after cardiac procedures: An updated meta-analysis. Pacing Clin Electrophysiol. 2020 Aug;43(8):856-865. doi: 10.1111/pace.14008. Epub 2020 Jul 20. PMID 32638389
- [Background] Atti V, Turagam MK, Garg J, Alratroot A, Abela GS, Rayamajhi S, Lakkireddy D. Efficacy and safety of figure-of-eight suture versus manual pressure for venous access closure: a systematic review and meta-analysis. J Interv Card Electrophysiol. 2020 Apr;57(3):379-385. doi: 10.1007/s10840-019-00547-6. Epub 2019 Apr 18. PMID 31001767
- [Background] Jensen CJ, Schnur M, Lask S, Attanasio P, Gotzmann M, Kara K, Hanefeld C, Mugge A, Wutzler A. Feasibility of the Figure-of-8-Suture as Venous Closure in Interventional Electrophysiology: One Strategy for All? Int J Med Sci. 2020 Apr 6;17(7):965-969. doi: 10.7150/ijms.42593. eCollection 2020. PMID 32308550